CLINICAL TRIAL: NCT00016861
Title: Pediatric Phase I and Pharmacokinetic Study of Irinotecan
Brief Title: Irinotecan in Treating Children With Refractory or Progressive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Children's Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TCCC-H-6957; CDR0000068568 (Registry Identifier: PDQ (Physician Data Query)); TCCC-GCRC-0654; NCI-V01-1654
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2004-11

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of irinotecan in treating children who have refractory or progressive solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of irinotecan in children with refractory or progressive solid tumors.
* Determine the pharmacokinetics of this drug and its metabolites (SN-38, SN-38G, and APC) administered with and without concurrent anticonvulsants in this patient population.
* Determine the benefit this drug offers this patient population.

OUTLINE: This is a dose-escalation, multicenter study. Patients are accrued into stratum 1 initially and into stratum 2 if stratum 1 closes due to dose-limiting toxicity of myelosuppression or diarrhea. Patients on anticonvulsants will be accrued into stratum 3 and must meet the eligibility criteria for the stratum that is open (stratum 1 or stratum 2). (Stratum 1 closed as of 2002-09-15).

Patients receive irinotecan IV over 90 minutes weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) with and without anticonvulsants is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: Approximately 20-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor refractory to standard therapy or for which no known effective therapy exists

  * Brain tumors eligible

    * Histologic verification waived for brain stem gliomas
* Evaluable disease
* No bone marrow involvement

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* Karnofsky 50-100% (over age 10)
* Lansky 50-100% (age 10 and under)

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGPT less than 5 times normal

Renal:

* Creatinine normal OR
* Glomerular filtration rate at least 70 mL/min

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 months since prior autologous bone marrow transplantation (BMT) (not including stem cell rescue after high-dose chemotherapy)
* At least 1 week since prior growth factors
* No prior BMT with total body irradiation (stratum I)
* No prior BMT with or without total body irradiation (stratum 2)
* No prior allogeneic BMT (all strata)
* No concurrent sargramostim (GM-CSF)
* No other concurrent prophylactic growth factor support during the first course of therapy

Chemotherapy:

* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* No prior irinotecan
* No more than 2 prior multi-agent chemotherapy regimens (stratum 2)
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent dexamethasone allowed if on stable or decreasing dose for at least 2 weeks prior to study

Radiotherapy:

* At least 6 months since prior craniospinal radiotherapy or radiotherapy to 50% or more of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* No prior central axis radiotherapy, pelvic radiotherapy, and/or total abdominal radiotherapy (stratum 2)

Surgery:

* Not specified

Other:

* Recovered from all prior therapy
* No other concurrent investigational agents
* Concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, phenobarbital, carbamazepine) allowed if on stable dose for at least 2 weeks prior to study (stratum 3)
* Concurrent valproic acid allowed if combined with another enzyme inducing anticonvulsant drug (stratum 3)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-09; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Blaney, MD, Study Chair — Texas Children's Cancer Center
Locations (1):
- Texas Children's Cancer Center, Houston, Texas, United States